CLINICAL TRIAL: NCT05925036
Title: Novel Cellular Therapy for the Treatment of Pain Associated With Chronic Pancreatitis
Acronym: MSCPainRelief
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NURP-003-22F; I01CX002516 (NIH)
Record Dates: First submitted 2023-06-20; First posted 2023-06-29 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pancreatitis; Chronic Pain
Keywords: Mesenchymal stem cells (MSCs); Chronic pancreatitis; Pain relief; Pancreas dysfunction; Fibrosis
MeSH Terms: conditions — Pancreatitis, Chronic; Chronic Pain; Fibrosis

STUDY DESIGN:
Intervention Model Description: This is a phase 1, randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability of a single intravenous infusion of autologous bone marrow-derived mesenchymal stromal cells in subjects with painful chronic pancreatitis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Experimental Cohort (Experimental): MSC
  Interventions: Drug: Mesenchymal stem cells
- Validation Cohort (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mesenchymal stem cells — Autologous bone marrow derived MSCs
  Other Names: MSCs
  Arms: Experimental Cohort
Other: Placebo — Controls
  Other Names: Control
  Arms: Validation Cohort

SUMMARY:
The goal of this clinical trial is to test whether adult stem cells, called mesenchymal stem cells (MSCs) collected from the patient's bone marrow can help reduce pain caused by chronic pancreatitis and improve pancreatic function.

DETAILED DESCRIPTION:
Chronic pain affects approximately 50 million U.S. adults and disproportionally impacts about 20 million veterans; 1 in 3 Veterans have been diagnosed with a condition related to chronic pain. There is also a significant interaction between chronic pain, post-traumatic stress disorder (PTSD), and persistent post-concussive syndromes common to the veteran population. The opioids that are prescribed to treat chronic pain are often ineffective and are associated with a significantly increased risk of misuse, addiction, diversion, overdose, and death. Unconventional treatment options that can effectively manage pain and avoid or reduce opioid addiction in Veterans are of significant clinical importance to VA healthcare. Given the high morbidity and mortality attributable to pain therapy, not to mention the staggering medical cost, it is vital to the VA healthcare mission to explore novel strategies to treat chronic pain effectively. Chronic pancreatitis (CP) is an inflammatory disease characterized by pancreatic inflammation, fibrosis, and abdominal pain. CP subjects often suffer extreme pain, which often leads to opioid addiction. In our animal models, the investigators show a linkage between inflammatory increases in neuropeptides and pain. In humans, the investigators have more specific pain measurements to explore the link between inflammation, neuropeptides, and neuropathic pain measurement as impacted by a novel therapeutic.

Mesenchymal stromal cells (MSCs) are adult stem cells that can be harvested and expanded for therapy. MSC therapy represents a promising new intervention as increasing evidence demonstrates that MSC therapy can effectively target several injury pathways in a variety of fibroinflammatory diseases and can reduce pain while suppressing inflammation, something that most pharmacological interventions cannot accomplish.

Rationale of the study: Because MSCs are a novel therapy that my improve chronic pancreatitis pain in animal models and improve chronic pain in other human disease states, these cells are worthy of study. Specifically, the investigators propose a pilot phase 1 crossover study design in which MSCs or placebo are prospectively given to CP subjects with pain outcomes measured. This phase 1 study will inform future study designs and may lead to MSCs as a standard of care if they are safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years old, male or female
* Definite chronic pancreatitis M-ANNHEIM criteria (Tsimmerman Ia, 2008) One or more of the following are required:
* Pancreatic calcifications
* Moderate or marked ductal lesions
* Marked and persistent exocrine insufficiency defined as pancreatic steatorrhea markedly reduced by enzyme supplementation
* Typical histology of an adequate histological specimen
* Patients who are diagnosed with painful CP for more than 6 months may be constant or may have been waxing and waning/remitting.
* Baseline Izbicki pain score > 30 (Dworkin et al., 2005)
* Stable dose of opioids for the past 30 days

Exclusion Criteria:

* Acute pancreatitis per 2012 revised Atlanta criteria (23) within the last 30 days oThe revised Atlanta classification requires that two or more of the following criteria be met for the diagnosis of acute pancreatitis: (a) abdominal pain suggestive of pancreatitis, (b) serum amylase or lipase level greater than three times the upper normal value, or (c) characteristic imaging findings.
* Chronic pain syndromes other than pancreatitis that require daily use of opioids in the past 30 days.
* Hemoglobin of <8.0g/dL, EGFR<60 ml/min, AST or ALT >2 times upper limit of normal, Bilirubin > 1.5 mg/dl unless the subject has confirmed Gilbert syndrome., Platelets <100,000/microliter, HbA1c >10%
* Congestive Heart Failure NYHA class >1
* History of Malignancy except for in situ malignancies that have been surgically treated and basal cell skin cancers
* Evidence of active infection using current antibiotics or with Hepatitis B, C, or HIV
* Known intravenous contrast allergy causing anaphylaxis
* Any subject who has had an ongoing alcohol abuse and/or illegal drug dependencies within the past six months.
* Any subject who has received an investigational drug or device within 30 days before randomization or who is expected to receive an investigational drug or device during this study.
* Patients with planned endoscopic or surgical intervention, surgical resection or needle drainage of pancreatic structures in the next 6 months.
* Subjects with infected pancreatic pseudocysts or pancreatic walled-off necrotic areas at the time of consent
* Females who are pregnant or women of childbearing potential (WOCBP) and males with female partners of childbearing potential who are not willing to use adequate contraception during the study
* Breastfeeding females
* Subject unwilling to follow the protocol and assessment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Izbicki pain score (M6 vs. Baseline) | 6 month
  Change in pain as measured by Izbicki pain scores

SECONDARY OUTCOMES:
Change in pancreatic volume measured by blinded scoring of MRI | Screening, 6 months and 12 months
  Pancreas volume change
Change in opioid use as measured in average daily morphine equivalents. | Screening, 6 and 12 months
  Average Daily morphine Equivalent.
Change in quality of life | Screening, 6 and 12 months
  Quality of life to be measured by Promise-29-v 2.1
Change in M-Manheim Severity Index absolute score | Screening, 6 and 12 months
  Severity of Index absolute scores

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun N Wang, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No